CLINICAL TRIAL: NCT03848273
Title: Clinical Diagnostic Criteria of Forecasting Epileptic Seizures in Stroke Patients
Brief Title: Post Stroke Epileptic Seizures Risk Forecast
Acronym: POSTER-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lviv National Medical University (Other)
Responsible Party: Principal Investigator, Andriy Kuzminskyy, Assistant of professor, Lviv National Medical University
Other Study IDs: LNMU-FPGE-Neuro-POSTER-1
Record Dates: First submitted 2019-01-23; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Stroke; Post Stroke Seizure; Post Stroke Epilepsy
Keywords: stroke; epilepsy; seizure; EEG
MeSH Terms: conditions — Stroke; Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ischemic: questionnaire, physical-neurological examination, labor investigations, EEG
- Hemorrhagic: questionnaire, physical-neurological examination, labor investigations, EEG
- Control: questionnaire, physical-neurological examination, labor investigations, EEG

SUMMARY:
Improve the effectiveness of treatment and prognosis in patients with cerebrovascular accident by early detection of the risk of developing epileptic seizures.

ELIGIBILITY:
Inclusion Criteria:

* informed consent to participate in the study signed by the patient / relative of the patient / the legal representative of the patient
* age over 18 years
* stroke, confirmed by neuroimaging
* light to moderate stroke (score on National Institutes of Health Stroke Scale).

Exclusion Criteria:

* recanalization therapy
* previous epileptic seizures and history of epilepsy
* psychiatric diseases in history
* previous stroke
* traumatic brain injury
* brain tumors.
* inflammatory and infectious diseases
* decompensated physical illness.
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient of Lviv Clinical Emergency Hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-02-20 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
First epileptic seizure | 1 year
  Patient's dairy will be used to assess this outcome measure.

SECONDARY OUTCOMES:
Longest seizure-free period | 1 year
  Patient's dairy will be used to assess this outcome measure.

OTHER OUTCOMES:
Death | 1 year
  Coroner report will be used to assess this outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Anzhelika Payenok, MD, DrMedSc, Prof, Study Chair — Danylo Halytsky Lviv National Medical University
Locations (1):
- Danylo Halytsky Lviv National Medical University, Lviv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided